CLINICAL TRIAL: NCT02603666
Title: Elastography of the Liver in Cystic Fibrosis Patients. Diagnostic and Prognostic Aspects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ferenc Karpati, MD, PhD, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010/1957/31/3
Record Dates: First submitted 2015-05-04; First posted 2015-11-13 (Estimated); Results first posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-11

CONDITIONS: Cystic Fibrosis; Liver Fibrosis
Keywords: cystic fibrosis; elastography; liver biopsy
MeSH Terms: conditions — Cystic Fibrosis; Liver Cirrhosis | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elastography (Other): Fibroscan elastography device for evaluation of liver disease in CF patients.
  Interventions: Device: Fibroscan

INTERVENTIONS:
Device: Fibroscan — Ultrasound by specific wavelength developed for elastography, repeated measures according to the manufacturer's instructions.
  Other Names: Elastography

SUMMARY:
The aim of the study is to find CF patients at risk for cystic fibrosis related liver disease (CFLD). Comparison of ultrasound by two modalities and biochemical markers with histological evaluation of liver biopsy if present.

DETAILED DESCRIPTION:
There are 209 CF patients attending Stockholm Cystic Fibrosis Center (January 2010). All up till 15 years of age are screened for liver disease annually by ultrasound (US) and also by biochemical markers. Ultrasound is performed every third year over 15 years of age in patients without CFLD, while all of them with diagnosed CFLD are continued to be investigated annually. Biochemical markers are controlled at least once every year in all CF patients. Elastography of the liver will be planned together with the investigations of the annual follow up, in an optimal clinical status. If either US or elastography of the liver indicates liver disease or progress of the already existing pathological changes, a liver biopsy will be performed according to routine procedure at Stockholm CF Centre. Also, historical data of liver biopsies and biochemical investigations will be considered in the study.

Elastography of the liver will be performed by Fibroscan device, with transducers for children and adults, respectively.

Clinical importance Liver US investigations in CF patients have important implications but are difficult to standardize in a routine clinical setting. Elastography may have an advantage in the evaluation of early fibrosis with clinical importance in pursuing diagnostics and intensifying treatment. A significant group (up to 25 %) of CF patients may be helped by this novel method. Including histological data, accuracy of elastography in CF patients may be improved. Further details of the importance of fatty acid status in CF may be elucidated.

ELIGIBILITY:
Inclusion Criteria:

* Verified cystic fibrosis

Exclusion Criteria:

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ferenc Karpati, MD, PhD, Principal Investigator — Stockholm CF Center, Karolinska University Hospital

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatient department, between 04/Feb/2012 and 04/Apr/2014
Period: Overall Study
Arm/Group | Elastography
Started | 130
Completed | 130
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Elastography
Number analyzed (Participants) | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 57
  Between 18 and 65 years | 71
  >=65 years | 2
Gender [Count of Participants; unit: Participants]
  Female | 73
  Male | 57
Region of Enrollment [Number; unit: participants] — Stockholm Cystic Fibrosis Center, Sweden Prospective inclusion
  participants
    Sweden | 130

OUTCOME MEASURES:

1. Primary Outcome: Elastographic Value in kPa Measured by Fibroscan
Description: Elastographic values given in kPa by Fibroscan. All patients undergo elastographic measurement of the liver and ultrasound of the liver. The grade of fibrosis is to be established by setting the cut-off for cystic fibrosis patients.
Time Frame: Within 28 days in connection with their annual evaluation at a single point of time
Measure: Mean (95% Confidence Interval); unit: kPa
Arm/Group | Elastography
Number analyzed (Participants) | 130
kPa | 4.7 [4.3 to 5]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Elastography
Serious Adverse Events (participants affected / at risk) | 0/130
Other Adverse Events (participants affected / at risk) | 0/130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No